CLINICAL TRIAL: NCT04233580
Title: Characterization of AmnioExcel Plus in Two Treatment Paradigms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Larry Lavery, Professor and Director of Research, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1527
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Weekly AmnioEXCEL+ group (Active Comparator): AmnioEXCEL+ will be applied weekly at study visits
  Interventions: Device: Amnio Excel + weekly
- PRN AmnioEXCEL+ group (Active Comparator): AmnioEXCEL+ will be applied maximum every 2 weeks (PRN, in the case that the wound requires debridement at a visit not intended for AE+ application, the wound will be treated as SOC)
  Interventions: Device: Amnio Excel + max every 2 weeks

INTERVENTIONS:
Device: Amnio Excel + weekly — Amnio Excel + weekly
  Arms: Weekly AmnioEXCEL+ group
Device: Amnio Excel + max every 2 weeks — Amnio Excel + max every 2 weeks
  Arms: PRN AmnioEXCEL+ group

SUMMARY:
The Investigators plan to evaluate healing in two cohorts of patients with diabetic foot wounds (n=20) that receive optimal treatment including serial wound debridement and off-loading with a boot or postop shoe and AmnioEXCEL+. In one cohort, AmnioEXCEL+ will be applied weekly at study visits and in the second cohort, AmnioEXCEL+ will be applied maximum every 2 weeks (PRN, in the case that the wound requires debridement at a visit not intended for AE+ application, the wound will be treated as SOC). In addition, the Investigators will collect data on other potential confounding factors that could affect healing such as antibiotic, anti-fungal and anti-infective medications, tobacco, comorbidities, diabetes control, infection, perfusion, and activity. Wound healing, including wound size and adverse events will be evaluated.

DETAILED DESCRIPTION:
Study Procedures:

Collection of Demographic data, medical/social history Collection of medications1 Ankle Brachial Index2 Wound debridement3 (standard of care procedure) Imaging with eKare4 Hyperspectral Imaging Application of study product

1. Only collect antibiotics, anti-fungal and anti-infective medications.
2. ABI (with toe pressure) can be done at screening or baseline.
3. Once wound is healed, wound debridement will not be done at weekly visits.
4. Once wound is healed, eKare will not be done at weekly visits.
5. EOS will occur on the date the subject is healed. *Screening and Visit 1 may be done on the same day.

Screening and Enrollment*:

* Review and sign the Informed Consent and HIPAA Authorization
* Review the inclusion and exclusion criteria

If the subject qualifies for the study, they will participate in the following procedures (weekly visits, +/-4 days):

Visit 1*:

* Demographics (such as age, gender, race or ethnicity)
* Past Medical History, Social History, Medications documented.
* Labs documented as SOC within 6mo of initial visit
* ABI with toe pressures2
* Wound debridement
* eKare wound measurement
* Hyperspectral Imaging
* Randomization
* Application of AmnioEXCEL+
* Source documentation
* Stipend disbursement

Visits 2 through 6:

* Wound debridement3
* eKare wound measurement4
* Hyperspectral imaging
* Application of AmnioEXCEL+ per cohort assignment
* Source documentation
* Stipend disbursement

Visit 7:

* Medications documented
* Wound debridement3
* eKare wound measurement4
* Hyperspectral imaging
* Application of AmnioEXCEL+ per cohort assignment
* Source documentation
* Stipend disbursement

Visits 8-11:

* Wound debridement3
* eKare wound measurement4
* Hyperspectral Imaging
* Application of AmnioEXCEL+ per cohort assignment
* Source documentation
* Stipend disbursement

Visit 12:

* Wound debridement3
* eKare wound measurement4
* Source documentation
* Stipend disbursement

End of Study (EOS) Visit 5:

* Medications documented
* Wound debridement3
* eKare wound measurement4
* Source documentation
* Subject exit from study

ELIGIBILITY:
Criteria for Inclusion of Subjects:

* 21-90 years of age
* Able to provide informed consent
* Chronic foot ulceration below the ankle - persistent for >30 days but <6 months

Criteria for Exclusion of Subjects:

* <21 or >90 years of age
* Unable to provide informed consent
* History of poor compliance in the opinion of the investigator
* Gangrene
* Untreated osteomyelitis
* Widespread malignancy
* Active alcohol or substance abuse such as cocaine, heroin, or methamphetamines that in the opinion of the investigator will impact the subject's participation in the study
* Pregnancy

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weekly AmnioEXCEL+ Group | PRN AmnioEXCEL+ Group
Started | 20 | 20
Completed | 15 | 16
Not Completed | 5 | 4
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly AmnioEXCEL+ Group | PRN AmnioEXCEL+ Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (15.3) | 57.6 (9.8) | 58.43 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 15 | 13 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.2 (7.8) | 32.3 (5.0) | 32.3 (6.6)
Neuropathy [Count of Participants; unit: Participants] | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Healed
Description: Number of participants whose wounds healed during the study timeframe. Reported as dichotomous yes/no.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly AmnioEXCEL+ Group | PRN AmnioEXCEL+ Group
Number analyzed (Participants) | 20 | 20
Participants | 6 | 10

2. Secondary Outcome: Wound Volume
Description: Wound volume measured by camera which performs a 3D measurement and calculates the volume at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cubic centimeters
Arm/Group | Weekly AmnioEXCEL+ Group | PRN AmnioEXCEL+ Group
Number analyzed (Participants) | 20 | 20
cubic centimeters | 1.2 (3.27) | 0.53 (1.44)

3. Secondary Outcome: Wound Area
Description: Wound measured by camera which performs a 3D measurement and calculates the area at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | Weekly AmnioEXCEL+ Group | PRN AmnioEXCEL+ Group
Number analyzed (Participants) | 20 | 20
square centimeters | 3.98 (4.87) | 3.15 (4.05)

4. Secondary Outcome: Tissue Oxygenation (StO2) of the Dorsal Foot
Description: Tissue oxygenation measured by hyperspectral imaging camera at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Weekly AmnioEXCEL+ Group | PRN AmnioEXCEL+ Group
Number analyzed (Participants) | 20 | 20
percentage of oxygen saturation | 65.89 (15.41) | 65.70 (9.31)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Weekly AmnioEXCEL+ Group | PRN AmnioEXCEL+ Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 6/20 | 5/20
Other Adverse Events (participants affected / at risk) | 9/20 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly AmnioEXCEL+ Group (N=20) | PRN AmnioEXCEL+ Group (N=20)
Below knee amputation (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Infection (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Trauma to foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ulcer worsening (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abrasion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly AmnioEXCEL+ Group (N=20) | PRN AmnioEXCEL+ Group (N=20)
New ulcer development (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Infection (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was limited due to Covid-19 pandemic. Occasional missed visits occurred when patients were quarantined and not allowed to present to clinic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04233580/Prot_SAP_000.pdf